CLINICAL TRIAL: NCT00939211
Title: A Double-blind, Double-dummy, Placebo-controlled, Randomised, Multi-centre, 5-way Cross-over, Single-dose Study to Investigate the Local and Systemic Effects of Inhaled AZD9164 Compared to Tiotropium in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: The Study Will Evaluate the Effect of AZD9164 in Patients With Chronic Obstructive Pulmonary Disease
Acronym: LaCrossE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Carin Jorup, MD/MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1882C00003
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Results first posted 2011-08-05 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease (COPD); efficacy; safety; inhalation; long-acting muscarinic receptor antagonist (LAMA)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — AZD9164; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- AZD9164 100 mcg First, then Placebo for Spririva (Experimental): 1 x AZD9164 solution for inhalation through nebulisation 100 mcg (lung deposited dose) + 1 x placebo for Spiriva dry powder for inhalation
  Interventions: Drug: AZD9164; Drug: Placebo
- AZD9164 400 mcg First, then Placebo for Spiriva (Experimental): 1 x AZD9164 solution for inhalation through nebulisation 400 mcg (lung deposited dose) + 1 x placebo for Spiriva dry powder for inhalation
  Interventions: Drug: AZD9164; Drug: Placebo
- AZD9164 1200 mcg First, then Placebo for Spiriva (Experimental): 1 x AZD9164 solution for inhalation through nebulisation 1200 mcg (lung deposited dose) + 1 x placebo for Spiriva dry powder for inhalation
  Interventions: Drug: AZD9164; Drug: Placebo
- Spiriva 18 mcg First, then Placebo for AZD9164 (Active Comparator): 1 x Spiriva dry powder for inhalation 18 mcg + 1 x placebo for AZD9164 (sodium chloride)
  Interventions: Drug: Tiotropium; Drug: Placebo
- Placebo for Spiriva First, then Placebo for AZD9164 (Placebo Comparator): 1 x placebo Spiriva dry powder for inhalation + 1 x placebo for AZD9164 (sodium chloride)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9164 — Solution for inhalation through nebulization, single dose
  Arms: AZD9164 100 mcg First, then Placebo for Spririva; AZD9164 1200 mcg First, then Placebo for Spiriva; AZD9164 400 mcg First, then Placebo for Spiriva
Drug: Tiotropium — Dry powder for inhalation, single dose
  Other Names: Spiriva
  Arms: Spiriva 18 mcg First, then Placebo for AZD9164
Drug: Placebo — Placebo

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic respiratory condition with deteriorating lung function over the years. Patients with COPD experience symptoms of shortness of breath, cough and sputum production. This study is to assess the treatment effects after inhalation of three different single doses of AZD9164 (100, 400 and 1200 mcg) and one single dose of tiotropium (18 mcg). One dose of placebo will be given as comparator. 25 patients are to participate in the study and all will be recruited in Sweden. Each patient will visit the study doctor 9 times during the study, whereof 5 visits will be overnight visits. All examinations, treatment and the follow-up is free of charge.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of COPD
* FEV1 40 - 80% of the predicted normal value (post-bronchodilator) and post- bronchodilator FEV1/FVC < 70%

Exclusion Criteria:

* Any clinically relevant abnormal findings at screening examinations
* Any clinically significant disease or disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leif Bjermer, Prof, MD, PhD, Principal Investigator — University Hospital in Lund, Sweden
Locations (3):
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Luleå
  - Research Site, Lund

REFERENCES:
- [Derived] Bjermer L, Bengtsson T, Jorup C, Lotvall J. Local and systemic effects of inhaled AZD9164 compared with tiotropium in patients with COPD. Respir Med. 2013 Jan;107(1):84-90. doi: 10.1016/j.rmed.2012.09.014. Epub 2012 Oct 23. PMID 23098686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study has been performed at four centers in Sweden. The first subject entered the study on 23 June 2009 and the last subject completed the study on 6 November 2009.
Period: AZD9164 100 Mcg First, Then Placebo
Arm/Group | Entire Study Population
Started | 28 (Cross-over study)
Completed | 28
Not Completed | 0
Period: AZD9164 400 Mcg First, Then Placebo
Arm/Group | Entire Study Population
Started | 28
Completed | 28
Not Completed | 0
Period: AZD9164 1200 Mcg First, Then Placebo
Arm/Group | Entire Study Population
Started | 28
Completed | 28
Not Completed | 0
Period: Spiriva 18 Mcg First, Then Placebo
Arm/Group | Entire Study Population
Started | 28
Completed | 28
Not Completed | 0
Period: Placebo
Arm/Group | Entire Study Population
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Number of Baseline Participants
Number analyzed (Participants) | 28
Age Continuous [Mean (Full Range); unit: years] | 64.2 [51 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1), Peak Effect Within 0 - 24 Hours Post-dose
Description: Maximum FEV1 value
Time Frame: 0, 15 min, 30 min, 60 min, 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, 14 h, 18 h, 22 h, 24 h
Measure: Mean (Standard Deviation); unit: L
Groups:
- AZD9164 100 Mcg First, Then Placebo for Spiriva: 1 x AZD9164 solution for inhalation through nebulisation 100 mcg (lung deposited dose) + 1 x placebo for Spiriva dry powder for inhalation
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
L | 1.71 (0.36) | 1.79 (0.39) | 1.72 (0.39) | 1.71 (0.35) | 1.63 (0.41)

2. Primary Outcome: Forced Expiratory Volume in One Second (FEV1), Average Effect Over 22 - 26 Hours Post-dose
Description: Trough FEV1 value
Time Frame: 22 h, 24 h, 26 h
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
L | 1.58 (0.38) | 1.63 (0.38) | 1.62 (0.38) | 1.57 (0.35) | 1.52 (0.39)

3. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1), Average Effect Over 0 - 24 Hours Post Dose
Description: Average FEV1 value
Time Frame: 0, 15 min, 30 min, 60 min, 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, 14 h, 18 h, 22 h, 24 h
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
L | 1.57 (0.36) | 1.63 (0.39) | 1.56 (0.38) | 1.58 (0.35) | 1.50 (0.40)

4. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1), Effect at 15 Minutes Post-dose
Description: 15 min FEV1 value
Time Frame: 15 min
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
L | 1.42 (0.38) | 1.30 (0.42) | 1.25 (0.44) | 1.55 (0.36) | 1.49 (0.42)

5. Secondary Outcome: Systolic Blood Pressure, Average Effect Over 0 - 4 Hours Post-dose
Description: Average systolic blood pressure value
Time Frame: 0, 30 min, 2 h, 4 h
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
mmHg | 125.5 (15.6) | 127.9 (14.8) | 127.3 (14.9) | 128.0 (13.3) | 126.5 (16.6)

6. Secondary Outcome: Diastolic Blood Pressure, Average Effect Over 0 - 4 Hours Post-dose
Description: Average diastolic blood pressure value
Time Frame: 0, 30 min, 2 h, 4 h
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
mmHg | 73.1 (7.9) | 75.6 (8.2) | 74.2 (6.7) | 74.8 (6.2) | 73.5 (8.6)

7. Secondary Outcome: Pulse, Average Effect Over 0 - 4 Hours Post-dose
Description: Average pulse value
Time Frame: 0, 30 min, 2 h, 4 h
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
bpm | 61.1 (7.6) | 62.9 (7.1) | 64.8 (8.0) | 60.2 (7.6) | 61.3 (7.5)

8. Secondary Outcome: Heart Rate, Average Effect Over 0 - 4 Hours Post-dose
Description: Average heart rate value
Time Frame: 0, 30 min, 2 h, 4 h
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
bpm | 61.0 (6.9) | 62.8 (7.8) | 65.2 (7.4) | 61.1 (7.4) | 61.3 (7.4)

9. Secondary Outcome: QTcF, Average Effect Over 0 - 4 Hours Post-dose
Description: Average QTcF value
Time Frame: 0, 30 min, 2 h, 4 h
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28
ms | 400 (23.1) | 399 (25.8) | 396 (25.0) | 401 (26.8) | 398 (23.1)

10. Secondary Outcome: Plasma AZD9164 Cmax
Description: Maximum plasma concentration of AZD9164
Time Frame: 0, 5 min, 15 min, 30 min, 60 min, 90 min, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h
Measure: Geometric Mean (Full Range); unit: nmol/L
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Number analyzed (Participants) | 27 | 28 | 28 | 0 | 0
nmol/L | 0.529 [0.24 to 1.55] | 3.629 [1.31 to 13.9] | 20.02 [6.15 to 70.2] |  |

11. Secondary Outcome: Plasma AZD9164 AUC0-24
Description: Area under the AZD9164 plasma concentration curve
Time Frame: 0, 5 min, 15 min, 30 min, 60 min, 90 min, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h
Measure: Geometric Mean (Full Range); unit: nmol*h/L
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Number analyzed (Participants) | 27 | 28 | 28 | 0 | 0
nmol*h/L | 2.90 [1.2 to 16.2] | 15.2 [6.9 to 66.8] | 58.1 [21.8 to 217] |  |

ADVERSE EVENTS:
Arm/Group | AZD9164 100 Mcg First, Then Placebo for Spiriva | AZD9164 400 Mcg First, Then Placebo for Spiriva | AZD9164 1200 Mcg First, Then Placebo for Spiriva | Spiriva 18 Mcg First, Then Placebo for AZD9164 | Placebo for Spiriva First, Then Placebo for AZD9164
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 4/28 | 15/28 | 27/28 | 2/28 | 3/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD9164 100 Mcg First, Then Placebo for Spiriva (N=28) | AZD9164 400 Mcg First, Then Placebo for Spiriva (N=28) | AZD9164 1200 Mcg First, Then Placebo for Spiriva (N=28) | Spiriva 18 Mcg First, Then Placebo for AZD9164 (N=28) | Placebo for Spiriva First, Then Placebo for AZD9164 (N=28)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 18 | 1 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 8 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 7 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 2 | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 3 | 0 | 0 | 2
Chest Discomfort (General disorders) | 0 | 2 | 4 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 2 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AZ for review at least 60 days in advance of submission for publication. Investigators in multicenter (MC) studies agree to postpone MC publications until the earlier of the date of the first AZ-authorized MC publication or a period up to 18 months from study completion at all sites. AZ has the right to request delays: up to 60 days for confidential information, and an additional 90 days to protect intellectual property.